CLINICAL TRIAL: NCT00641459
Title: Behavioral and Psychological Symptoms of Dementia (BPSD) in Taiwan - An Observational Study
Brief Title: A Study on Behavioral and Psychological Symptoms of Dementia
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CR014665
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Dementia
Keywords: Behavioral and Psychological Symptoms of Dementia; BPSD; NPI; CGI; MMSE
MeSH Terms: conditions — Dementia; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001
  Interventions: Other: Observational BPSD treatment study

INTERVENTIONS:
Other: Observational BPSD treatment study — Observational BPSD treatment study

SUMMARY:
The purpose of this observational study is to obtain the current status of patients with Behavioral and Psychological Symptoms of Dementia. This study is also expected to further provide insight into the evolution of behavioral and psychotic symptoms and its relationship with treatment as well as severity of cognitive declines in a naturalistic setting.

DETAILED DESCRIPTION:
This is an observational, prospective, multi-center study to obtain information about the symptoms and treatment received for patients with behavioral and psychological symptoms of dementia (BPSD). Patients must first meet eligibility criteria and sign informed consent. Patient treatment will be based upon investigator opinion. The following parameters will be assessed: patient's characteristics, Clinical Global Impression (CGI) score, Neuropsychiatric Inventory (NPI), and Minimal Mental Status Examination (MMSE). Each patient will be observed for 12 weeks. Medication dosing regimen will be flexible throughout the study and is based on patient response and investigator judgment. During the study observation period, all patients will attend clinic visits for the subsequent 12 weeks (visit 2 to 3) as is the usual clinical practice. Patients can visit clinics on additional dates as needed or by request. At the pre-planned clinic visits, CGI score, NPI, vital signs, reports of adverse events, drug information, and MMSE score (visit 3) will be recorded. This is an observational study and no study drug is administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of dementia according to DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) criteria
* Patients meet one of the following types of Dementia: Dementia of the Alzheimer's Type (AD), Vascular Dementia (VaD), Dementia of Lewy Body (DLB), Parkinson's Disease Dementia (PDD)
* Patients have one or more active symptoms of Behavioral and Psychological Symptoms of Dementia (BPSD) on Neuropsychiatric Inventory (NPI) and have not received treatment with antipsychotics, mood stabilizers, or antidepressants within 1 month prior to study entry
* Patients are with caregiver(s) who can give appropriate information about the patients and can assist with the assessment during the study
* Patients (or a legally acceptable representative) have signed the informed consent form

Exclusion Criteria:

* Patients with concurrent other primary major psychiatric disorders (such as Schizophrenia or Bipolar disorder)
* Patients with history of severe allergies or multiple adverse drug reactions
* Patients with history or current symptoms of tardive dyskinesia
* Patients with history of neuroleptic malignant syndrome (NMS)
* Patients who participated in a clinical trial of any investigational drug within 1 month (30 days) prior to study entry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males or females with diagnosis of dementia according to DSM-IV criteria
Sampling Method: Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
This observational study is to obtain the characteristics, distribution of symptoms, and treatment of patients, including dosages and duration, among subjects with behavioral and psychological symptoms of dementia (BPDS) in a naturalistic setting. | 12 weeks

SECONDARY OUTCOMES:
CGI (Clinical Global Impression) scores in week 4, week 12, versus in Baseline. | 12 weeks
MMSE (Minimal Mental Status Examination) scores in week 12 versus in Baseline. | 12 weeks
NPI (Neuropsychiatric Inventory) scores in week 4, week 12, versus in Baseline. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd